CLINICAL TRIAL: NCT03497520
Title: The Effect of Asymmetric Spinal Stabilization Exercise on Scoliosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-1701/377-305
Record Dates: First submitted 2018-03-29; First posted 2018-04-13 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Scoliosis Idiopathic
Keywords: surface EMG; cobb angle; exercise; Spinal Curvatures
MeSH Terms: conditions — Motor Activity; Spinal Curvatures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- scoliosis patients (Experimental): scoliosis patients who have cobb angle over 10 degree perform asymmetric spinal stabilization exercise
  Interventions: Behavioral: asymmetric spinal stabilization exercise

INTERVENTIONS:
Behavioral: asymmetric spinal stabilization exercise — The patients were educated to strengthening weakness side of spinal muscle, as asymmetric spinal stabilization exercise(ASSE)
  * before teach ASSE, the investigators will evaluate Cobb angle, Apical vertebral rotation in Adam's test, surface EMG, Scoliosis Research Society-22(SRS-22) quastionnaire for evaluation of scoliosis severity
  * after perform ASSE, the investigators will evaluate Cobb angle, Apical vertebral rotation in Adam's test, surface EMG, Scoliosis Research Society-22(SRS-22) quastionnaire for evaluation of scoliosis severity

SUMMARY:
The purpose of this study is to evaluate the effect of asymmetric spinal stabilization exercise on scoliosis

DETAILED DESCRIPTION:
* Design: Prospective study
* Setting: hospital rehabilitation department
* Intervention: Participants are educated asymmetric spinal stabilization exercise along scoliosis curve patterns, including the location of apex and the direction of convexity. After performing asymmetric spinal stabilization exercise, participants are compared the main outcome measures.
* Main outcome measures: Cobb angle, Apical vertebral rotation in Adam's test, surface EMG, Scoliosis Research Society-22(SRS-22) quastionnaire

ELIGIBILITY:
Inclusion Criteria:

* who have idiopathic scoliosis, showing at Cobb's angle over 10 degrees on X-ray

Exclusion Criteria:

* Patients who underwent spinal surgery
* Patients with spinal scoliosis due to cerebral palsy, muscle paralysis, polio, congenital spinal abnormalities
* Patients observed with Cobb's angle less than 10 degrees, over 40 degrees
* Patients complaining of acute low back pain

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
cobb angle | through study completion, an average of 6 months
  measure lateral curve of vertebra on spine x-ray AP view
Apical vertebral rotation | through study completion, an average of 1 year
  angle of trunk rotation in Adam's test
surface electromyography | through study completion, an average of 6 months
  surface muscle contraction of bilateral spinal muscle on T7, T12, L3

SECONDARY OUTCOMES:
Scoliosis Research Society-22(SRS-22) quastionnaire | through study completion, an average of 1 year
  five different factors (pain, self-image/appearance, function/activity, mental health, and satisfaction with management, 5 = best; 1 = worst)the minimum and maximum score range is from 5 to 25

CONTACTS AND LOCATIONS:
Overall Officials: Jusuk Ryu, M.D. PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided